CLINICAL TRIAL: NCT06923709
Title: Beneficial Effect of Amiloride on Progression of Chronic Kidney Disease
Acronym: A-CKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EUCT: 2022-500692-31-00; 2022-500692-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-02; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease(CKD); Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Amiloride

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double blinded, placebo controlled, crossover study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiloride (Experimental): Amiloride 5mg twice daily for 7 days followed by 2-3 weeks of washout and then placebo twice daily for 7 days
  Interventions: Drug: amiloride
- Placebo (Placebo Comparator): Placebo twice daily for 7 days followed by 2-3 weeks of washout and then Amilorid 5 mg twice daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: amiloride — 5mg twice daily for 7 days
  Arms: Amiloride
Drug: Placebo — 1 tablet twice daily for 7 days
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blinded crossover trial testing the effects of amiloride in patients with chronic kidney disease (CKD) and proteinuria.

In CKD with proteinuria, there is aberrant filtration of serine proteases and complement precursors into the tubular lumen. The interaction of these factors leads to proinflammatory complement activation, which may promote inflammation, opsonization, and formation of the membrane-attack complex, causing cell injury.

With the aim of preserving kidney function, reducing cardiovascular morbidity, and delaying renal replacement therapy in CKD, this study tests whether amiloride (10 mg/day) protects the filtration barrier, lowers albuminuria, and mitigates kidney inflammation through urokinase inhibition, independent of blood pressure effects.

Participants are randomized to receive amiloride (10 mg/day) or placebo for one week, with a 2-3-week washout period in between. Blood and urine samples are collected before and after each treatment period. Additionally, ECG, body composition measurements, blood pressure, and body weight are monitored.

The primary outcome measures are urinary C3a, soluble C5-9 (sTCC/MAC), and kidney injury biomarkers KIM-1 and NGAL. Secondary endpoints include the urinary albumin/creatinine ratio, protein/creatinine ratio, and blood pressure.

DETAILED DESCRIPTION:
Please refer to the protocol

ELIGIBILITY:
Inclusion criteria

Participants are eligible to be included in the study, only if all the following criteria apply:

1. Participant must be 18 years of age including at the time of signing the informed consent.
2. A clinical diagnosis of chronic kidney disease and:

   1. eGFR ≥ 25 mL/min/1.73m2 and < 60mL/ min/1.73m2 at screening
   2. UACR of ≥ 300mg/g at screening
3. Participants must be on stable antihypertensive treatment 2 weeks before start of study drug and throughout study duration.
4. Office blood pressure at screening meeting (visit 1), > 110/60mmHg and < 150/90mmHg. If BP > 150/90mmHg at visit 1, screening phase can be prolonged to 4 weeks#.
5. Capable of giving signed informed consent.
6. Women with childbearing potential* can only be included if a pregnancy test is negative at the screening visit. Moreover, women should be using contraception during the study.

   * If the office blood pressure varies by approximately ±10 mmHg and is deemed acceptable by the investigator, the participant can be included.

     * Women are considered of childbearing potential following menarche and until becoming post-menopausal (12 consecutive months without a menstrual period) unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy or bilateral oophorectomy (According to the Clinical Trial Facilitation Group, 2014-09-15).

Exclusion criteria

Participants are excluded from the study is any of the following criteria apply:

1. Treatment with amiloride alone or in combination or use of other types of K-sparing diuretics, MR antagonists (Spironolactone, eplerenone, finerenone)
2. Ongoing cancer treatment
3. Treatment with immunosuppressive therapy within 6 months prior to screening
4. History of organ transplantation
5. Evidence of current infection (CRP> 50 and temperature > 38◦C)
6. History of unstable or rapidly progressing renal disease (eGFR decreasing > 5ml/min/1.73m2 the last 2 months)
7. Severe hepatic insufficiency classified as Child-Pugh C
8. Patients on hypertension treatment who is not on stable antihypertensive treatment 2 weeks before start of study drug.
9. Pregnancy or breastfeeding participants
10. Congestive heart failure NYHA class IV, unstable or acute congestive heart failure.
11. Recent cardiovascular events in a patient:

    1. Less than two months post coronary artery revascularization.
    2. Acute stroke or TIA within two months prior to screening
    3. Acute coronary syndrome within two months prior to screening
12. Patients who, in the judgement of the investigator may be at risk for dehydration.
13. Known hypersensitivity to the study treatment (active substance or excipients)
14. Known hypersensitivity to resonium
15. Addison´s disease
16. Gastric bypass operation
17. Participation in other interventional trials
18. Lactose intolerance
19. Plasma potassium >4.9 mmol/l at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Urine-C3a (ng/ml) | Measured before (day one) and after (day 8) each treatment period
  Urine-C3a is measured in spot urine samples and expressed as u-C3a/creatinine (µg/g) to account for the dilution factor.
Urine C5-9-sTCC/MAC (U/ml) | Measured before (day one) and after (day 8) each treatment period
  Membrane Attack Complex (MAC) of the complement system, specifically targeting the C5 to C9 proteins. u-C5-9 is measured in spot urine samples and expressed as u-C5-9/creatinine U/µmol to account for the dilution factor.
Kidney Injury Molecule-1 (KIM-1) pg/ml | Measured before (day one) and after (day 8) each treatment period
  KIM-1 is a protein that serves as a biomarker used particularly in the context of kidney injury
Neutrophil Gelatinase-Associated Lipocalin (NGAL) (pg/mL) | Measured before and after each treatment period
  NGAL is a protein associated with neutrophils used as a biomarker in the context of kidney injury.

SECONDARY OUTCOMES:
Urine albumin/creatinin ratio (mg/g) | Measured before (day one) and after (day 8) each treatment period
  In spot urine samples, albumin and creatinin are measured
Urine protein/creatinin ratio | Measured before (day one) and after (day 8) each treatment period
  In spot urine samples, albumin and creatinin are measured
Home blood pressure (mmHg) | Measured before (day one) and after (day 8) each treatment period
  Home blood pressure are measured according to standard guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No